CLINICAL TRIAL: NCT05288439
Title: Neuroimaging Biomarkers of Impaired Neurocognitive Functioning After Cranial Proton Beam Radiotherapy For Treatment of Brain Tumors In Pediatric Patients
Brief Title: A Study of How Proton Beam Radiotherapy (PBRT) Affects Brain Function and Quality of Life in Children and Young Adults Undergoing Treatment for a Brain Tumor
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-061
Record Dates: First submitted 2022-03-08; First posted 2022-03-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Brain Tumor; Metastatic Brain Tumor
Keywords: Proton Beam Radiotherapy (PBRT); Cognitive battery assessment; Quality of life assessment
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: This prospective, cross-sectional, pilot clinical trial will incorporate rs-fcMRI and a full post- PBRT cognitive battery including quality of life assessment for pediatric patients using a multidisciplinary team.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients (Experimental): A full neurocognitive battery with quality-of-life assessment will be conducted and an rs-fcMRI sequence will be added to the brain MRI performed as standard of care follow-up between 3-5 months post-PBRT.
  Interventions: Diagnostic Test: Resting-state functional connectivity MRI; Other: Neurocognitive battery with quality-of-life assessment
- healthy matched controls (Experimental): Healthy participants will be asked to complete the MRI scan and undergo neurocognitive assessment.
  Interventions: Diagnostic Test: Resting-state functional connectivity MRI; Other: Neurocognitive battery with quality-of-life assessment

INTERVENTIONS:
Diagnostic Test: Resting-state functional connectivity MRI — participants will undergo functional MRI
Other: Neurocognitive battery with quality-of-life assessment — Cognitive and quality of life assessments performed by a trained neuropsychologist

SUMMARY:
The researchers are doing this study to find out if there are differences in the resting state brain networks of children and young adults (ages 6-25) after treatment with proton beam radiation therapy (PBRT). The researchers will use resting state functional connectivity magnetic resonance imagining (rs-fcMRI) scanning to detect these differences. The researchers will also check for differences in participants' thinking and quality of life through a cognitive assessment and a questionnaire. Both people undergoing PBRT for a brain tumor and healthy people will take part in this study so that the researchers can compare the brain networks (connections in the brain that are involved in certain function, such as memory or attention), thinking patterns, and quality of life of these two groups of participants.

The study researchers think that rs-fcMRI scans may be an effective way to look at the brain networks after treatment with PBRT and see if this treatment causes differences in those networks, including damage to the brain (neurotoxicity). rs-fcMRI scans take images when a patient is in a resting state, which means the patient is not performing a task or thinking about anything in particular.

This study will provide valuable information about how PBRT affects brain networks, thinking (cognitive) abilities, and quality of life in children and young adults. The study results may have an impact on future treatment approaches for brain cancer and the use of PBRT in children and young adults.

ELIGIBILITY:
Inclusion Criteria:

Patients Treated for Brain Tumors:

* The patient has been diagnosed with a primary or metastatic brain tumor
* The patient has been recommended to receive cranial PBRT for a primary or metastatic brain tumor
* The patient is between the ages of 6 through 25 at time of consent
* As per medical record or patient report (based on prior tolerance of MRI), the participant is able to tolerate MRI without sedation (i.e., general anesthesia). Patients will take medications as prescribed or directed by the patient's physician. If in accordance with their prescribed regimen, agents that may impact the CNS, such as benzodiazepines and/or antihistamines, should be avoided on the day of imaging and neurocognitive assessment.

Healthy Control Participants:

* The control has no major medical illness, as determined by medical interview by study physician
* As per parent report, the control is between the ages of 6 through 25 at time of consent
* As per parent report, the control is able to tolerate an MRI without sedation (i.e., general anesthesia). Participants should only take medications as prescribed or directed by their physician. They should not take additional medications, such as antihistamines, for the purpose of tolerating MR imaging.

Exclusion Criteria:

* As per self or parent report, the participant has completed any portion of the neuropsychological battery used in this study within the last year.
* As per medical record or self or parent report, there is an existing diagnosis of intellectual disability and/or prior IQ testing that documents Full Scale IQ standard score <70 at baseline.
* As per medical record, there is an existing diagnosis of psychiatric disorder or untreated mood disturbance, prior stroke or intracranial hemorrhage, or neurodegenerative disease.
* The participant has an MRI contraindication (e.g., implanted ferromagnetic devices, claustrophobia) as per radiology clinical operating procedures.
* As per self or parent report, non-fluency in English language as demonstrated by current educational placement in a non-English-speaking classroom setting.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
differences in the resting state brain networks of children and young adults | 1 year
  A single rs-fcMRI sequence will be added to the MRI performed as standard of care follow-up 3-5 months after completion of cranial PBRT in pediatric patients treated for brain tumors to assess for early post-PBRT network disruption.
  Using resting state functional connectivity magnetic resonance imagining (rs-fcMRI) scanning to detect these differences.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Holodny, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm